CLINICAL TRIAL: NCT01466894
Title: A Randomized, Double-Blind, Placebo-Controlled Dosing, Safety and Efficacy Study of IMM 124-E (Bovine Colostrum) for Patients With Nonalcoholic Steatohepatitis
Brief Title: Safety and Efficacy Study of IMM 124-E (Bovine Colostrum) for Patients With Nonalcoholic Steatohepatitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor administrative decision
Sponsor: Immuron Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NASH-Immuron-002
Record Dates: First submitted 2011-11-02; First posted 2011-11-08 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: Nonalcoholic fatty liver disease; NAFLD; Fatty liver; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- IMM 124-E high dose (Experimental): IMM 124-E 3600 mg per day
  Interventions: Biological: IMM 124-E
- IMM 124-E low dose (Experimental): IMM 124-E 1800 mg per day
  Interventions: Biological: IMM 124-E
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: IMM 124-E — Tablets orally twice a day for 24 weeks
  Other Names: Bovine colostrum powder
  Arms: IMM 124-E high dose; IMM 124-E low dose
Biological: Placebo — Tablets orally twice daily for 24 weeks
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, placebo-controlled, double-blind, dose-selection, multiple dose administration study comprising three groups, with up to 40 patients in each active treatment and placebo group. Patients with biopsy proven nonalcoholic steatohepatitis (NASH) and elevated liver enzymes will be randomized to undergo a liver MRI scan and to receive Imm 124-E or placebo for 24 weeks. During this period, patients will be followed for clinical and laboratory effects. At the end of 24 weeks of treatment, patients will undergo a second liver MRI scan. Patients will be followed for an additional 4 weeks for safety after completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 to 75 years (inclusive)
* Subjects with biopsy proven NASH (NAS ≥ 4) within one year prior to screening
* Elevated liver enzymes at screening and at least once within past 6 months (ALT > 30 women, ALT > 40 men)
* Normal or only slightly impaired synthetic liver function (serum albumin >3.5gm%, INR 0.8-1.5)
* BMI 18 to 40 (inclusive)
* Subjects able to adhere to the visit schedule and protocol requirements and be available to complete the study
* Women of child bearing potential must be using adequate contraception

Exclusion Criteria:

* Cow milk allergy or lactose intolerance
* Excessive alcohol use (Women > 20 grams/day, Men > 40 grams/day).
* Current treatment with Insulin or Incretins
* Decompensated liver disease
* Other or concomitant cause of liver disease (viral hepatitis, autoimmune liver disease, metabolic liver disease, vascular liver disease)
* Subjects who known to be HIV positive
* Subjects who have undergone surgery within the last 3 months
* Subjects who have had a prior gastrointestinal surgery
* Subjects who have a history of Inflammatory Bowel Disease
* Subjects who are receiving an elemental diet or parenteral nutrition
* Subjects with an infectious, immune-mediated or active malignant disease (during the last 3 months)
* Subjects with known clinically significant systemic disease
* Subjects treated with other anti-NASH therapy(s) - thiazolidinediones, vitamin E, SAM-e, betaine, milk thistle, gemfibrozil, anti-TNF therapies and probiotics) - within 3 months of the liver biopsy
* Subjects who have been treated with any type of immune modulatory drug, including systemic steroids or NSAIDs, within the last 3 months
* Subjects who have received either Immuron, 6-MP, Methotrexate, Cyclosporine, anti-TNF alpha therapies (Infliximab, Adalimumab, Etanercept) or anti-integrin therapies (namixilab) within the past 12 months
* Known history of drug or alcohol abuse, including positive urinary drugs of abuse screen at the screening visit
* Subjects who are pregnant as confirmed on screening test
* Any acute medical situation (e.g. acute infection) within 48 hours of study start that is considered of significance by the Principal Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Safety outcome | 28 weeks
  No unexpected treatment related SAEs throughout the participation period and the follow up period

SECONDARY OUTCOMES:
MRI liver fat quantitation | Baseline and 24 weeks
  Improvement in MRI fat quantification as determined by a decrease in the fat content by 5% or more from baseline to week 24
ALT levels | Baseline and 24 weeks
  Normalization of alanine aminotransferase levels in patients with NASH from baseline to week 24
Liver enzyme improvement | Baseline and 24 weeks
  Improvement in liver enzymes by 20% from baseline from baseline to week 24
Lipid profile | Baseline and 24 weeks
  Improvement in lipid profile by 20% from baseline from baseline to week 24
HbA1c | Baseline and 24 weeks
  Improvement in HBA1c by 0.5 % from baseline from baseline to week 24